CLINICAL TRIAL: NCT07054866
Title: Rural Autistic Individuals - Supporting Expression
Acronym: RAISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Nadezhda Modyanova, Assistant Research Professor, Montana State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-73
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Autism Disorder; Language Development Disorders; ADHD; Typical Development; Rural Health; Children; Neuroimaging; Eye Tracking; EEG; fNIRS
MeSH Terms: conditions — Autistic Disorder; Language Development Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Language Evaluation (Experimental)
  Interventions: Behavioral: Speech-Gesture combinations

INTERVENTIONS:
Behavioral: Speech-Gesture combinations — this is a pretest, test, posttest evaluation of language comprehension with and without gestures, to see if gestures can improve language comprehension

SUMMARY:
This research study investigates how hand gestures can support language comprehension and communication skills of hearing speaking, non-speaking, and/or minimally verbal individuals with Autism Spectrum Disorders (ASD), who are especially disadvantaged by the lack of accessible services in their rural communities. Individuals with other cognitive profiles, including Developmental Language Disorder (DLD), ADHD, Dyslexia, and others are welcome too. The study uses methods of eye tracking and recording of brain activity to understand how hand gestures adapted from signs from American Sign Language, such as [cry], can promote successful understanding of words like "cry". The overarching goal is to help families effectively utilize gestures to support communication with their children.

DETAILED DESCRIPTION:
The investigators are researching how hand gestures and signs from American Sign Language influence language comprehension, and whether gestures/signs can support communication in children and adults with social and language impairments.

The investigators use non-invasive brain imaging methods (skin-contact only). One is EEG - electroencephalography - which records electrical brain activity on scale of milliseconds. Another is fNIRS (functional near infrared spectroscopy) which shines infrared light through scalp and measures blood flow to the brain areas which are more active during a task. The researchers employ a protocol that uses both neuroimaging methods at the same time. This involves wearing a cloth helmet, and having a lot of wires attached to the surface of the helmet. The EEG wires need gel to be put into hair to pick up the brain signal.

For psychological measurements, there are three rounds of tasks. One set of tasks about language and gestures happens as passive viewing of a computer screen with pictures of common objects and videos of a person gesturing and speaking. For example, see a picture for a dog, and hear "dog", and see gesture for "dog". There's no response required here.

Another set of tasks is in picture books to evaluate language comprehension and IQ for solving puzzles, if the participant has capacity to engage with the picture books, if not - that's optional.

Third task is 3-5 questionnaires for adults/caregivers about demographics, diagnoses (if any), experience with services, and autism, ADHD, and communication.

All together the study takes at least 2-3 hours of research time per participant, plus breaks. Both children and adults are welcome participate.

ELIGIBILITY:
Inclusion Criteria:

* 1.1 Confirmed (preferably) or suspected diagnosis of ASD (autism spectrum disorder), or a receptive language impairment (i.e., difficulties with comprehension, Developmental Language Disorder), or both. Additional diagnoses, including ADHD (Attention Deficit and Hyperactivity Disorder), are acceptable. Siblings and cousins of these individuals are also welcome.

OR 1.2 No diagnoses of ASD or DLD for unrelated control typically-developing participants.

2. Normal hearing and normal vision (or corrected to normal with glasses or contacts).

3. Ages 2+. 4. English as the dominant language of caregivers. 5. Caregivers who self-identify as living in a rural area. 6. The ability to verbally or physically respond is optional.

Exclusion Criteria:

* 1. Poor hearing. 2. Inborn or acquired brain damage.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
EEG/ERP brain response | from Enrollment to completion of study protocol within 3 months
  In a pretest-test-postest set up, the researchers measure participants' EEG/ERP (electroencephalography/event related potentials) signals in microvolts ﬁrst prior to exposure to gestures, just with visual animations and auditory words; then the investigators expose participants to visual gestures with auditory words; and ﬁnally participants are exposed to animations and auditory words again, to see if gestures contributed to any changes in EEG/ERP.

SECONDARY OUTCOMES:
fNIRS brain response | from enrollment to completion of protocol within 3 months
  In a pretest-test-postest set up, the researchers measure participants' brain activation via blood flow response using fNIRS (functional near infrared spectroscopy). The investigators identify whether language or non-language brain areas are activated during animation, speech, or gestures.

CONTACTS AND LOCATIONS:
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data, including language and cognitive evaluations, along with EEG and fNIRS.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after peer-reviewed publications from this study are made public
Access Criteria: appropriate data use agreements will need to be put in place

REFERENCES:
- [Background] Poplin, M., Ma, J., Aviles Zuniga, T., Modyanova, N., Johnson, E., McCrory, B. (March 2025). Using Electroencephalography to Understand Learning Engagement with User-Centered Human-Computer Interaction in a Multimodal Online Learning Environment. Annual Conference of the Institute of Industrial and Systems Engineers (IISE).
- [Background] Modyanova, N.N., Bolton, A. P., Storrusten, C., & McCrory, B. (2024). Improving Language Comprehension via Hand Gestures in Children with Autism Spectrum Disorders and/or Language Impairment in Rural Montana. Proceedings of the International Symposium on Human Factors and Ergonomics in Health Care, 13(1), 191-196. https://doi.org/10.1177/2327857924131012
- See also: Biomedical Innovation for Research and Development Hub supports the implementation of this study — https://coe.montana.edu/bioredhub/